CLINICAL TRIAL: NCT05884268
Title: Evaluating Safety and Tolerability of Venlafaxine for Postoperative Pain of Laparoscopic Cholecystectomy
Brief Title: Venlafaxine for Postoperative Pain of Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Principal investigator-Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6-2023
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Cholecystectomy (Active Comparator)
  Interventions: Drug: Venlafaxine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Venlafaxine — Patients scheduled for elective LC will receive 150 mg venlafaxine before surgery
  Arms: Laparoscopic Cholecystectomy
Drug: Placebo — Patients scheduled for elective LC will receive placebo venlafaxine before surgery
  Arms: Control

SUMMARY:
Recent studies on the impact of perioperative venlafaxine for treatment of acute postoperative pain have yielded positive outcomes . The aim of the present study is to investigate the role of perioperative venlafaxine on the management of postoperative pain in patients undergoing LC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who are scheduled to undergo elective LC

Exclusion Criteria:

1- Patients with acute pancreatitis 2. Patients undergoing chronic pain treatment 3. Patients who received analgesics or sedatives 24 h before scheduled surgery 3. Patients had alcohol or drug addiction 4. Severe hepatic and renal dysfunction 5. Previous allergic response to duloxetine 6. Pregnancy and lactation 7. Patients with communication problems, cognitive dysfunction, or psychological disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain between the two groups using visual analogue score (VAS) | 24 Hours postoperative
  pain will be assessed using visual analogue score (VAS) 0-100 mm (0 indicated no pain, 100 denoted the most severe pain)
  pain will be assessed using visual analogue score (VAS) 0-100 mm (0 indicated no pain, 100 denoted the most severe pain)

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24 Hours postoperative
  will be assessed using PONV scale a 4-point scale: none (0): no nausea, vomiting, and retching; mild (1): happened once; moderate (2): happened 2-3 times; and severe (3): continuous or more than three times.

IPD SHARING:
Plan to Share IPD: Undecided